CLINICAL TRIAL: NCT00002351
Title: An Open-Labeled, Multiple Dose, Multicenter Study to Investigate the Safety, Tolerability, and Plasma Concentration Profile of L-735,524 Capsules in HIV-Seropositive Older Children and Adolescent Patients
Brief Title: A Study of L-735,524 in HIV-Positive Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246A; 026-01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; HIV Protease Inhibitors; Indinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Indinavir

INTERVENTIONS:
Drug: Indinavir sulfate

SUMMARY:
To evaluate the safety, tolerability, and plasma concentration profiles of indinavir sulfate ( MK-639; Crixivan ) in HIV-seropositive older children and adolescents. To compare the plasma concentration profile after the initial dose with data from a historical group of adults. To obtain preliminary data on antiviral activity of MK-639.

DETAILED DESCRIPTION:
Patients receive MK-639 for 14 and one-third days. Repeat plasma samples are collected up to 8 hours following the first and last dose. Urine samples are collected on days 1 and 5.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity.
* No active opportunistic infection within the past 30 days, other than superficial candidiasis of the oral cavity or vagina.
* Body surface area at least 1.0 sqm.
* Consent of parent or guardian.

Prior Medication:

Allowed:

* Aerosolized pentamidine.
* Topical antifungals.
* TMP / SMX.
* AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant hepatic disease including HBsAg or hepatitis C positivity.
* Significant neurologic disease such as loss of intellectual ability, motor deficits, or seizure disorder.
* Significant cardiac disease including dysrhythmia or cardiomyopathy.
* Significant medical condition or laboratory abnormality that may pose additional risk to patient on study or confound the results.
* Has a social situation that may interfere with study participation.

Concurrent Medication:

Excluded:

* Oral contraceptives.

Patients with the following prior conditions are excluded:

* History of serious allergic drug reactions.
* History of significant cardiac disease.
* Participation on another clinical trial within the past 4 weeks.
* Donated blood within the past 4 weeks.

Prior Medication:

Excluded within the past 4 weeks:

* Hematopoietic growth factors.

Excluded within the past 2 weeks:

* Antiretroviral agent other than zidovudine.
* Oral contraceptives.
* Prophylaxis for opportunistic infections, other than aerosolized pentamidine, topical antifungals, and TMP/SMX.
* Any other medication unless approved by Merck clinical monitor. Current illicit drug use.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Locations (1):
- Merck & Co Inc, Whitehouse Station, New Jersey, United States

REFERENCES:
- [Background] Mueller BU, Sleasman J, Nelson RP Jr, Smith S, Deutsch PJ, Ju W, Steinberg SM, Balis FM, Jarosinski PF, Brouwers P, Mistry G, Winchell G, Zwerski S, Sei S, Wood LV, Zeichner S, Pizzo PA. A phase I/II study of the protease inhibitor indinavir in children with HIV infection. Pediatrics. 1998 Jul;102(1 Pt 1):101-9. doi: 10.1542/peds.102.1.101. PMID 9651421